CLINICAL TRIAL: NCT02868203
Title: Optical Coherence tOmography Based Edge and In-stent Vascular Response After a Novel bioDegradable Polymer sIrolimus-eLuting Stent in patIents With Non-ST Elevation acuTe Coronary sYndrome (NSTE ACS)
Brief Title: OCT Based Edge and In-stent Vascular Response After Cordimax Stent in patIents With NSTE-ACS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ky20162025-1
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-05

CONDITIONS: Angina, Unstable; Non-ST-Segment Elevation Myocardial Infarction
MeSH Terms: conditions — Angina, Unstable | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OCT at 3 months (Active Comparator): OCT at 3 months and 12 OCT at 3 months
  Interventions: Device: OCT; Device: eLuting stent
- OCT at 6months (Active Comparator): OCT at 6 months and 12 OCT at 3 months
  Interventions: Device: OCT; Device: eLuting stent

INTERVENTIONS:
Device: OCT — OCT after stent implantation
Device: eLuting stent

SUMMARY:
This study evaluates the completeness of strut coverage and vessel wall response, at different time points (3-6-12 Months), following CordimaxTM stent implantation in patients with non-ST elevation acute coronary syndrome

DETAILED DESCRIPTION:
Major concerns were addressed to the delayed healing process of drug-eluting stents . To date no studies have detailed the in-vivo completeness of CordimaxTM stent coverage at different time points. The objective of this prospective study is to measure the completeness of strut coverage and vessel wall response (neointima disomogeneity, acquired late incomplete strut apposition) at different time points following CordimaxTM stent implantation, in patients with non-ST elevation acute coronary syndrome . Optical Coherence Tomography (OCT) that detects smaller degrees of stent strut coverage more accurately than IVUS will be used at different time points (3-6-12 Months)

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 and ≤ 75 years
2. Non-ST-segment elevation MI
3. Patient willing to comply with specified follow-up

5.Patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided written informed consent 6.Single or two de novo or non-stented restenotic lesion in a native coronary artery 7. Target lesion to be covered by a single stent of max 30 mm . Reference vessel diameter ≥2.25 to ≤ 4.0 mm by visual estimate 8. The vessel diameter should be measured after pre-dilation procedure and after intra-coronary nitroglycerin if spasm is suspected 9. Target lesion ≥70% stenosed by visual estimate

Exclusion Criteria:

1. Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure. Female patients of childbearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test
2. Impaired renal function or on dialysis
3. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3 or a WBC<3,000 cells/mm3
4. Patient has a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated
5. Patient requires low molecular weight heparin (LMWH) treatment postprocedure or has received a dose of LMWH ≤8 hours prior to index procedure
6. Patient has received any organ transplant or is on a waiting list for any organ transplant;
7. Patient has other medical illness or known history of substance abuse that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (<1 year)
8. Patient has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/ticlopidine, prasugrel, stainless steel alloy, sirolimus and/or contrast sensitivity that cannot be adequately pre-medicated
9. Patient has previously received murine therapeutic antibodies and exhibited sensitization through the production of Human Anti-Murine Antibodies
10. Patient presents with cardiogenic shock
11. Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion;
12. Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study
13. Currently participating in another investigational drug or device study or patient in inclusion in another investigational drug or device study during follow-up
14. Calcified target lesion(s) which cannot be successfully predilated
15. Target lesion has excessive tortuosity unsuitable for stent delivery and deployment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of uncovered and/or malapposed bioDegradable polymer sIrolimus-eLuting stent at 12 month after the implant, as measured by OCT | 12 month

IPD SHARING:
Plan to Share IPD: Yes